CLINICAL TRIAL: NCT05798026
Title: A Dose-escalation, Single-arm, Open-Label, Phase 1 Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of EU103 in an Advanced or Metastatic Solid Tumors Who Have Failed Standard Therapy
Brief Title: A Phase 1 Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of EU103 in Advanced or Metastatic Solid Tumors That Have Failed Standard Therapy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eutilex (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EU-CTS103-I-01
Record Dates: First submitted 2023-03-22; First posted 2023-04-04 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- EU103: Dose Escalation Cohort (Experimental): Participants with advanced solid tumors will receive EU103 intravenously once every 3 weeks (3 weeks = 1 cycle) with escalating doses starting from 1 milligrams per kilogram (mg/kg) for each cohort and increasing to 3, 6, 12 or 24 mg/kg until disease progression, unacceptable toxicities or death, withdrawal of consent, end of study, or physician's decision, whichever occurs first.
  Interventions: Drug: EU103
- EU103: Dose Escalation Cohort 1 (Experimental): 1 mg/kg
  Interventions: Drug: EU103
- EU103: Dose Escalation Cohort 2 (Experimental): 3 mg/kg
  Interventions: Drug: EU103
- EU103: Dose Escalation Cohort 3 (Experimental): 6 mg/kg
  Interventions: Drug: EU103
- EU103: Dose Escalation Cohort 4 (Experimental): 12 mg/kg
  Interventions: Drug: EU103
- EU103: Dose Escalation Cohort 5 (Experimental): 24 mg/kg
  Interventions: Drug: EU103
- Backfill cohort (Other): Additional subjects can be registered at doses confirmed to be safety
  Interventions: Drug: EU103

INTERVENTIONS:
Drug: EU103 — EU103 will be administered via intravenous infusion.

SUMMARY:
Phase 1 (dose escalation) of this study will evaluate:

The safety and tolerability of EU103 treatment are evaluated for patients with advanced or metastatic solid tumors who have failed standard therapy to determine the maximum tolerated dose and recommended Phase 2 dose.

And preliminary efficacy (tumor response), The pharmacokinetic characteristics are evaluated, and changes are investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males or females aged 18 years (or 19 years according to local regulatory requirements) or older at the time of obtaining written consent
2. Patients with histologically or cytologically confirmed unresectable advanced or metastatic solid tumors who have failed locally known standard therapies or are unable to apply any more standard therapies.
3. Patients with at least 1 measurable or non-measurable lesion per RECIST v1.1
4. Patients with an estimated survival of 3 months or longer, as determined by the investigator
5. Patients with ECOG PS 0-2
6. Patients with adequate bone marrow, liver, and renal functions at the time of screening

   * Absolute Neutrophil Count (ANC) ≥ 1,500 /μL
   * Platelet ≥ 100,000 /μL
   * Hemoglobin ≥ 9.0 g/dL (If the hemoglobin level of a patient is below 9.0 g/dL, he/she may be enrolled upon recovery to 9.0 g/dL or higher. However, blood transfusions performed in order to meet this criterion within 14 days before screening are not allowed.)
   * AST and/or ALT ≤ 2.5x ULN (≤ 5 x ULN if liver metastases are present)
   * Total bilirubin ≤ 1.5 x ULN (≤ 3 x ULN if liver metastases are present)
   * Serum creatinine ≤1.5 x ULN

     * However, if serum creatinine is >1.5 x ULN, Creatinine clearance (CrCl) ≥ 60 mL/min is allowed for enrollment.
   * PT (INR) ≤1.5 x ULN
7. Those who provide or can provide newly obtained tumor biopsies (preferred) or archived tumor tissue specimens during the screening period.

   In patients recruited to the dose escalation phase for DLT evaluation, provision of tumor tissue specimens is preferred but not required.

   Patients included in cohort reinforcement must agree to provide a tumor tissue specimen during the screening period and to undergo an additional biopsy in cycle 1 (before the start of cycle 2).

   If possible, cycle 1 (before cycle 2) biopsies should be obtained from the same organ site as the biopsy provided at screening to avoid heterogeneity related to tumor or metastatic sites.

   The neoplastic lesion to be used for a newly acquired biopsy should not be a target lesion unless there are no other suitable lesions, in which case only central needle (non-excisional/non-incisional) biopsy should be performed. It is allowed.

   Specimens from metastatic bone lesions are generally not accepted unless they have a significant soft tissue component. The amount of tumor specimen should be sufficient to allow exploratory biomarker analysis, preferably in the form of formalin-fixed paraffin-embedded blocks or slides.
8. For women of childbearing potential, the serum pregnancy test is negative
9. Women of childbearing potential or men who do not plan for pregnancy during the study and for 6 months after the last dose of investigational product and who agree to maintain the following clinically appropriate methods of contraception during the period

   * Hormonal contraceptive methods (such as subdermal implants, injections, oral contraceptives, etc.), intrauterine device (IUD) or Intra uterine system (IUS), sterilization surgery of the subject or the subject's partner (vasectomy, tubal ligation, etc.), double barrier methods (such as combined use of a cervical cap or a diaphragm with a male condom)
10. Patients who have given their written consent to voluntarily participate in this study

Exclusion Criteria:

1. Patients who have received prior anticancer therapy, monoclonal antibodies, chemotherapy, live vaccines, or other investigational products, or have a history of treatment with an investigational medical device within 4 weeks prior to the first dose of the investigational product
2. Patients who have not recovered (to Grade 1 or better, or the baseline level per NCI-CTCAE v5.0) from the adverse events (excluding alopecia) caused by prior anticancer therapy based on the start date of the first dose of the investigational product
3. Patients with a history of radiotherapy within 2 weeks prior to the investigational product administration Note. Subjects must have recovered from all radiation-related toxicities, not require corticosteroid use, and have no history of radiation pneumonitis. A 1-week recovery period is allowed for palliative radiotherapy (not more than 2 weeks of radiotherapy) for diseases other than the central nervous system (CNS) diseases.
4. Patients with a history of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonia, idiopathic pneumonia, or evidence of active pneumonia, or past history of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis requiring steroid treatment, or evidence of clinically active ILD
5. Patients with symptomatic ascites or pleural effusion Note. Enrollment is allowed if clinically stable after treatment for the condition (including thoracentesis or paracentesis for therapeutic purposes).
6. Patients with uncontrolled tumor-related pain (Patients with symptomatic lesions that can be treated with palliative radiotherapy [e.g., bone metastases or metastases causing nerve impingement] can be enrolled after treatment prior to screening).
7. Patients with known symptomatic, untreated, or actively progressing brain metastases and/or leptomeningeal disease
8. Patients who have had or currently have any of the following infections:

   * Individuals with a history of human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS) (However, patients with human immunodeficiency virus (HIV) who have no history of opportunistic infection and a CD4+ T cell (CD4+) count ≥350 cells/uL within 12 months prior to screening are allowed for enrollment)
   * Patients with active hepatitis B (However, those who have negative HBV titer based on the determination of the study site within 14 days prior to screening, have received antiviral therapy for at least 14 days prior to screening and are willing to maintain it throughout the study period are eligible for enrollment.)
   * Patients with active hepatitis C (However, if patients have completed antiviral treatment and their HCV viral load is negative based on the determination of the study site, they are eligible for enrollment.)
   * Patients with active infection accompanied by uncontrolled severe chronic infection or requiring treatment
9. Patients who have been diagnosed with a malignancy other than the indication in this study within 5 years prior to screening (However, patients who have been assessed as having complete response after treatment and have not relapsed within at least 3 years from the time of screening, or patients with non-melanoma skin cancer, in-situ disease, thyroid cancer, or borderline tumors are eligible for enrollment)
10. Patients with severe cardiac diseases clinically significant as determined by the investigator

    * Including but not limited to the following diseases: uncontrolled hypertension, congestive heart failure [NYHA Grade 2 or higher], ventricular arrhythmia, active ischemic heart disease, myocardial infarction within 1 year prior to screening, QTcF ≥ 450 ms (males) / ≥ 470 ms (females), or other cardiac diseases that, in the judgment of the investigator, preclude participation in this study.
11. Patients who are expected to require major surgery requiring general anesthesia within 4 weeks prior to administration of the investigational product or during the study
12. Patients who have received immunosuppressants within 2 weeks prior to the investigational product administration However, enrollment is allowed in the following cases: i) intranasal, inhaled, applied steroids or topical steroids; ii) prednisone less than 10 mg/day or equivalent dose of other corticosteroids; iii) steroids for prevention of hypersensitivity.
13. Patients who have received drugs targeting V-set and immunoglobulin domain containing 4 (VSIG4)
14. Patients with a history of hypersensitivity to the components of the investigational product or drugs in the same class (humanized/human monoclonal antibody treatments)
15. Pregnant women, lactating women, or those who are planning to become pregnant during this study period
16. Patients who are determined to be inappropriate for participation in this study as determined by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-08-08 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Event (AEs) and Serious Adverse Events (SAEs) and Adverse Events | Baseline up to 30 months
  Number of Participants With Adverse Event (AEs) and Serious Adverse Events (SAEs) and Adverse Events Leading to Discontinuation
Dose Limiting Toxicity (DLT) | At the end of Cycle 1 (Each cycle is of 21 Days)
  Number of Participants With Dose Limiting Toxicity (DLT)
Phase 1:Number of Participants With Clinically Significant Abnormalities in Laboratory Parameters | Time Frame: Baseline up to 24 months
  Laboratory assessments include hematology, serum chemistry, other blood tests, coagulation, and urine analysis. Number of participants with clinically significant abnormalities will be reported.
Number of participants with clinically significant abnormalities | Time Frame: Baseline up to 24 months
  Vital signs will include body temperature, pulse rate, and systolic and diastolic blood pressure measurements. Number of participants with clinically significant abnormalities will be reported.
Phase 1:Number of Participants With Clinically Significant Abnormalities in Physical Examination | Time Frame: Baseline up to 24 months
  Physical examination will include head, eyes, ears, nose and throat; heart; lungs; abdomen; skin; cervical and axillary lymph nodes; and neurological and musculoskeletal systems. Number of participants with clinically significant abnormalities will be reported.
Phase 1:Number of Participants With Clinically Significant Abnormalities in 12-lead Electrocardiogram (ECG)Physical Examination | Time Frame: Baseline up to 24 months
  ECG parameters included heart rhythm, pulse rate intervals, QRS, QT intervals, RR intervals and corrected QT(QTc) intervals. Number of participants with clinically significant abnormalities will be reported.
Phase 1:Production of anti-drug antibodies (ADAs) | Time Frame: Baseline up to 30 months
  The number of subjects, percentage, and Exact 95% confidence interval for subjects who are anti-drug antibody (ADA) positive at each measurement time point compared to before administration of investigational drugs are presented for each dose level.

SECONDARY OUTCOMES:
Phase 1:Objective response rate (ORR) | Time from first dose of study treatment assessed until disease progression, death, withdrawal of consent, physician's decision, start of new anticancer therapy, or end of study, whichever occurs first (approximately for 24 months)
  Proportion of subjects whose best overall response (BOR) is confirmed as complete response (CR) or partial response (PR)
Phase 1:Duration of response (DoR) | Time from first dose of study treatment assessed until disease progression, death, withdrawal of consent, physician's decision, start of new anticancer therapy, or end of study, whichever occurs first (approximately for 24 months)
  Time from achievement of tumor response (CR or PR) to the time of confirmed progressive disease (PD)
Phase 1:Disease control rate (DCR) | Time from first dose of study treatment assessed until disease progression, death, withdrawal of consent, physician's decision, start of new anticancer therapy, or end of study, whichever occurs first (approximately for 24 months)
  Proportion of subjects whose BOR is confirmed as CR, PR, or stable disease (SD: 6 weeks or longer)
Phase 1:Time to response (TTR) | Time from first dose of study treatment assessed until disease progression, death, withdrawal of consent, physician's decision, start of new anticancer therapy, or end of study, whichever occurs first (approximately for 24 months)
  Time from the date of the investigational product administration to the time of confirmed objective response (CR or PR)
Phase 1:Time to progression (TTP) | Time from first dose of study treatment assessed until disease progression, death, withdrawal of consent, physician's decision, start of new anticancer therapy, or end of study, whichever occurs first (approximately for 24 months)
  Time from the date of the investigational product administration to the time of PD
Phase 1:Progression-free survival (PFS) | Time from first dose of study treatment assessed until disease progression, death, withdrawal of consent, physician's decision, start of new anticancer therapy, or end of study, whichever occurs first (approximately for 24 months)
  Time from the date of the investigational product administration to the time of PD or death from any cause, whichever occurs first
Phase 1:Overall survival (OS) | Time from first dose of study treatment assessed until disease progression, death, withdrawal of consent, physician's decision, start of new anticancer therapy, or end of study, whichever occurs first (approximately for 24 months)
  Time from the date of the investigational product administration to death due to any cause

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Asan Medical Center, Seoul
  - Samsung Seoul Hospital, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No